CLINICAL TRIAL: NCT07120737
Title: Efficacy and Safety of Spectacle Lenses With Maximized Highly Aspherical Lenslets Target Technology (H.A.L.T. MAX) on High Myopia Control in Children and Adolescents: a Randomized Controlled Research
Brief Title: Efficacy and Safety of Spectacle Lenses With H.A.L.T. MAX Technology on High Myopia Control in Children and Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WS10422; IIT2024-019-AMD-01 (Other: Shanghai Eye Disease Prevention and Treatment Center)
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Myopia; High Myopia
Keywords: myopia; high myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: In a 2-year randomized controlled study, the intervention group wore H.A.L.T. MAX for at least 10 hours a day for 2 years. The control group will wear single vision lenses (SV) for at least 10 hours a day. In the first year (at 6-month follow-up), study participants in the control group with a spherical equivalent diopter change (SER) of ≥0.75 D will be switched to H.A.L.T. MAX lenses until the end of year 2. After entering year 2, all remaining control (SV) study participants will be replaced with H.A.L.T. MAX spectacles for at least 10 hours per day until the end of year 2. Only the study spectacles can be worn during the research study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): the intervention group wore H.A.L.T. MAX for at least 10 hours a day for 2 years.
  Interventions: Device: H.A.L.T. MAX spectacles
- The control group (No Intervention): The control group will wear single vision lenses (SV) for at least 10 hours a day. In the first year (at 6-month follow-up), study participants in the control group with a spherical equivalent diopter change (SER) of ≥0.75 D will be switched to H.A.L.T. MAX lenses until the end of year 2. After entering year 2, all remaining control (SV) study participants will be replaced with H.A.L.T. MAX spectacles for at least 10 hours per day until the end of year 2.

INTERVENTIONS:
Device: H.A.L.T. MAX spectacles — The Essilor® Stellest® 2.0 lens features a 2 times larger signal area, significantly enhancing the effect of slowing down myopia progression
  Arms: the intervention group

SUMMARY:
Children aged 7-14 years with high myopia were randomly assigned to a control group or an intervention group at a 1:1 ratio. The intervention group wore H.A.L.T. MAX lenses for at least 10 hours per day for 2 years, and the control group wore ordinary single-vision (SV) spectacles for at least 10 hours per day. At the 1-year follow-up examination (6-month visit), control subjects whose equivalent spherical diopter change (SER) was ≥0.75 D were switched to H.A.L.T. MAX lenses until the end of year 2. After entering year 2, all remaining control (SV) subjects will be replaced with H.A.L.T. MAX defofocus frames for at least 10 hours per day until the end of year 2. And continue to wear it for at least 10 hours per day. To evaluate the efficacy, safety and compliance of H.A.L.T. MAX lenses in delaying myopia progression in children with high myopia, and to provide a scientific basis for the formulation and practice of public health programs for delaying myopia progression and the risk of blindness and visual impairment caused by high myopia.

DETAILED DESCRIPTION:
In a 2-year randomized controlled study, the intervention group wear H.A.L.T. MAX spectacle lenses for more than 10 hours a day for 2 years. During the first year, the control group wore conventional single-vision (SV) spectacles for at least 10 hours per day. At the 6-month follow-up visit, if the spherical equivalent refraction (SER) change in the control group (SV) participants was ≥0.75 D, they were switched to H.A.L.T. MAX spectacle lenses until the end of the second year. In the second year, all remaining control group (SV) participants were transitioned to H.A.L.T. MAX defocus spectacle lenses and continued wearing them until the study concluded. To evaluate the efficacy, safety and compliance of H.A.L.T. MAX lenses for delaying myopia in children with high myopia, and to provide a scientific basis for the development of prevention strategies for children with high myopia.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, willing to follow the protocol, able to read and understand the information form and give free and informed consent (for parents/guardian of children subjects) and assent (for subjects aged 7-14 years old);
* 7-14 years old，regardless of sex;
* Spherical equivalent refraction (SE) after cyclopegia ≤ -5.00 D and ≥ -9.00D;
* Anisometropia and Astigmatism ≤2.50D;
* Best corrected distance visual acuity of at least 0.8 in both eyes;
* Willing to wear only the spectacles provided by the investigator for all days (>10 hours) during the study without additional interventions;
* Accept randomization;
* Able to sign the informed consent form with the accompaniment and understanding of parents or guardians.

Exclusion Criteria:

* Allergic or intolerant to cycloplegic drugs；
* Exclude children on high dose atropine (1%) or red light therapy；
* Any previous history of myopia control treatment in the previous 30 days, like low dose atropine, defocus spectacles, or thokeratology and acupuncture；
* History or presence of an ocular disease, strabismus or amblyopia or other binocular vision abnormalities, accommodation dysfunction, and cataract.；
* History of eye surgery；
* Ocular or systemic diseases that may be associated with myopia, such as Marfan syndrome, retinopathy of newborns, diabetes, etc；
* Anatomic or skin factors affecting the wearing of spectacles；
* Other conditions unsuitable for inclusion (patients with excessive expectations for the effect of the defocus spectacle lenses or desires to try other myopia interventions).

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
the proportion of change in SER of ≤ -0.75 (D) | at the end of 1-year
  the proportion of change in SER of ≤ -0.75 (D) at the end of 1-year in both groups

SECONDARY OUTCOMES:
The proportion of change in AL of ≥ 0.34 mm | at the end of 1-year
  The proportion of change in AL of ≥ 0.34 mm at the end of 1-year in both groups

OTHER OUTCOMES:
Adaptation outcome | at the end of 1-year
  visual quality, assessed by specify questionnaire.
Adverse events incidence | 1 year
  Number of participants with adverse events (e.g., headache, dizziness) attributed to lens wear.
Exploratory outcomes1 | at the end of 2-year
  Changes in SER and AL in the SVL switch over group in the second year.
Exploratory outcomes2 | at the end of 2-year
  Changes in choroidal thickness from baseline in the intervention and control group by OCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center (SEDPTC), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No